CLINICAL TRIAL: NCT06879548
Title: Bedside Assessment of Immune Function in Patients With Covid-19
Acronym: LITCOME
Status: Withdrawn | Type: Observational
Why Stopped: Study team moved
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 282113
Record Dates: First submitted 2021-04-10; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Covid19
Keywords: Immune; Neutrophil; Covid 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Covid-19 is a global pandemic causing unprecedented morbidity and mortality in the general population. It appears to have a greater effect on the elderly or those with underlying health problems but is not exclusively confined to these groups. As people age, particularly toward the end of their lives, the response of the immune system begins to drop away, an occurrence known as immunosenescence. It is known that there exist a group of people that do not respond to immune stimulation in a normal way but who may to observers be considered fit and healthy. The leukocyte immune test (LIT) relies upon the supramaximal stimulation of white cells outside of the body to determine their reactiveness when stimulated. It is intended to study patients admitted to Barts Health with diagnosed Covid-19. 4 ml blood will be taken of which 10microlitres will be used for the LIT. The remainder will be used for measurement of antibody levels previously associated with poor outcome following cardiac surgery. The patients will be followed up to see the proportion that progress to requirement for critical care, advanced ventilatory support, renal failure and in-hospital mortality. If a link can be established between a poor outcome following admission to hospital with Covid-19 and the immune response on admission, as predicted by means of the LIT, then it may enable better formulation of potential treatment strategies. Being able to measure at point of admission the responsiveness of someone's immune system may mean that treatment strategies such as the administration of passive immunization either via convalescent plasma or gammaglobulin will be better guided. If the LIT proves able to identify those people at risk of severe disease it may be able to identify individuals amongst healthcare workers that may benefit from passive immunisation or avoidance of high-risk exposure to Covid-19.

ELIGIBILITY:
Inclusion Criteria:

* Over 18y age Suspected diagnosis of Covid-19 Able to give written informed consent

Exclusion Criteria:

* Unwilling or unable to give consent Under 18years of age Suffering from other acute septic/infective illness other than Covid-19

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients passing through A&E with Covid-19 requiring admission to hospital without fulfilling the exclusion criteria will be potential recruits to the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-03-11 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Review point of care test of immune function at admission relate to progression of disease | From admission date to discharge date.
  Whether the result from a point of care test of immune function at admission relates to progression of disease requiring intensive care admission in hospitalised Covid-19 patients.

SECONDARY OUTCOMES:
Review LIT result at admission relate to requirement for respiratory support | Throughout patient hospital stay (admission date to discharge date).
  Whether the LIT result at admission relates to the requirement for respiratory support
Review LIT result at admission relate to requirement for renal replacement therapy | Throughout patient hospital stay (admission date to discharge date).
  Whether the LIT result at admission relates to the requirement for renal replacement therapy
Review LIT result at admission relate to length of admission | Throughout patient hospital stay (admission date to discharge date).
Review LIT result at admission relates to all cause in-hospital mortality | Throughout patient hospital stay (admission date to discharge date).
  Whether the LIT result at admission relates to all cause in-hospital mortality
Review the LIT result at admission relates to previously measured immune markers of associated with outcome, namely EndoCAb. | At 6 months
  Whether the LIT result at admission relates to previously measured immune markers of associated with outcome, namely EndoCAb.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Hamilton-Davies, Principal Investigator — Barts Health
Locations (1):
- Newham University Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided